CLINICAL TRIAL: NCT07373301
Title: Determination of the Protective Efficacy of the PvCS/Montanide ISA-51 Vaccine Formulation Against Controlled Infection With Plasmodium Vivax Sporozoites
Brief Title: Phase IIa/b Trial of PvCS/Montanide ISA-51 Malaria Vaccine in Adults in Chocó, Colombia
Acronym: PvCS/M51
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Malaria Vaccine and Drug Development Center (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2201-3
Record Dates: First submitted 2025-11-13; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Plasmodium Vivax Malaria; Plasmodium Vivax Infection; Malaria Prevention
Keywords: PvCS Vaccine; Plasmodium vivax; Malaria Vaccine; Montanide ISA-51; Controlled Human Malaria Infection; Malaria Prevention; Phase II Clinical Trial; Immunogenicity; Vaccine Efficacy; Colombia; Adult Volunteers
MeSH Terms: conditions — Malaria, Vivax

STUDY DESIGN:
Intervention Model Description: This study uses a randomized, double-blind, placebo-controlled, parallel-group design. Seventy-two healthy adults (18-50 years) from malaria-endemic areas of Chocó, Colombia, will be randomized 2:1 to receive PvCS/Montanide ISA-51 VG vaccine or placebo. Vaccinations will be given intramuscularly at 0, 2, and 4 months. One month after the final dose, all participants will undergo a controlled human malaria infection (CHMI) using Anopheles albimanus mosquitoes infected with Plasmodium vivax. Participants will be followed for infection, immune responses, and safety for up to 12 months
Who Masked: Participant, Investigator
Masking Description: Randomization and blinding procedures ensure that neither participants nor study staff involved in data collection or outcome assessment are aware of group allocation. Vaccine and placebo are identical in appearance and administration schedule.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Naïve Participants - PvCS/Montanide ISA-51 Vaccine (Experimental): Healthy adults with no prior malaria exposure will receive three intramuscular doses of the PvCS/Montanide ISA-51 VG vaccine at months 0, 2, and 4. The formulation contains a synthetic peptide representing the circumsporozoite protein (CS) of Plasmodium vivax combined with Montanide ISA-51 VG adjuvant. Participants will be monitored for safety and immune responses before undergoing controlled human malaria infection (CHMI) about one month after the final vaccination.
  Interventions: Biological: PvCS/Montanide ISA-51 VG Vaccine
- Naïve Participants - Placebo (Placebo Comparator): Healthy malaria-naïve adults will receive three intramuscular injections of placebo (adjuvant without PvCS antigen) on the same schedule as the vaccine arm (months 0, 2, and 4). Procedures for safety monitoring, blood sampling, and CHMI will be identical to those for the vaccine group. This arm serves as the negative control for efficacy and immunogenicity comparisons.
  Interventions: Biological: Placebo - Montanide ISA-51 VG Adjuvant Alone
- Semi-Immune Participants - PvCS/Montanide ISA-51 Vaccine (Experimental): Adults with prior natural exposure to malaria will receive three intramuscular doses of the PvCS/Montanide ISA-51 VG vaccine at months 0, 2, and 4. Safety and immune parameters will be assessed throughout the vaccination phase. Approximately one month after the final dose, participants will undergo CHMI with P. vivax to determine vaccine-induced protection in semi-immune individuals.
  Interventions: Biological: PvCS/Montanide ISA-51 VG Vaccine
- Semi-Immune Participants - Placebo (Placebo Comparator): Semi-immune adults will receive three intramuscular injections of placebo (adjuvant without PvCS antigen) following the same schedule as the vaccinated groups. Participants will undergo the same clinical, laboratory, and parasitological monitoring during vaccination and CHMI. This arm provides comparative data for evaluating vaccine safety and efficacy in semi-immune populations.
  Interventions: Biological: Placebo - Montanide ISA-51 VG Adjuvant Alone

INTERVENTIONS:
Biological: PvCS/Montanide ISA-51 VG Vaccine — The vaccine contains a synthetic peptide representing the central repeat and flanking regions of the Plasmodium vivax circumsporozoite (CS) protein, formulated with Montanide ISA-51 VG (Vaccine Grade), a water-in-oil adjuvant that enhances both antibody and T-cell responses. This formulation is distinct from other malaria vaccine candidates because it specifically targets P. vivax using a synthetic CS peptide antigen, rather than a recombinant protein or viral vector platform. Each 0.5-mL dose is administered intramuscularly in the deltoid at 0, 2, and 4 months. Participants will be closely monitored for safety, reactogenicity, and immunogenicity after each vaccination. Approximately one month after the final dose, volunteers will undergo a controlled human malaria infection (CHMI) via exposure to Anopheles albimanus mosquitoes infected with P. vivax sporozoites to assess protective efficacy.
  Other Names: PvCS Synthetic Peptide Vaccine; PvCS/ISA-51 VG
  Arms: Naïve Participants - PvCS/Montanide ISA-51 Vaccine; Semi-Immune Participants - PvCS/Montanide ISA-51 Vaccine
Biological: Placebo - Montanide ISA-51 VG Adjuvant Alone — The placebo consists of Montanide ISA-51 VG (Vaccine Grade) adjuvant without the Plasmodium vivax circumsporozoite (CS) peptide antigen. It is a sterile water-in-oil emulsion prepared and administered in the same manner as the investigational vaccine to maintain blinding. Each 0.5-mL dose is given intramuscularly in the deltoid at 0, 2, and 4 months. The placebo is visually indistinguishable from the vaccine and follows identical handling, storage, and administration procedures. Participants in the placebo group will undergo the same safety monitoring, blood sampling, and controlled human malaria infection (CHMI) one month after the final dose to allow direct comparison of efficacy, safety, and immune responses.
  Other Names: Naïve Participants - Placebo; Semi-Immune Participants - Placebo
  Arms: Naïve Participants - Placebo; Semi-Immune Participants - Placebo

SUMMARY:
This clinical study will evaluate an investigational malaria vaccine called PvCS/Montanide ISA-51 to determine whether it is safe and whether it can protect adults from infection with Plasmodium vivax, one of the main parasites that causes malaria. P. vivax malaria is common in tropical regions, including Colombia, and can lead to recurrent fever, anemia, and prolonged illness. Currently, no licensed vaccine effectively prevents P. vivax infection.

The investigational vaccine (PvCS) contains synthetic peptides derived from the circumsporozoite (CS) protein located on the surface of P. vivax sporozoites. The vaccine is formulated with the adjuvant Montanide ISA-51 to enhance the immune response. This study aims to assess the safety of the PvCS/Montanide ISA-51 formulation and to determine whether it can prevent malaria after controlled exposure to the parasite.

This is a Phase IIa/b, randomized, double-blind, placebo-controlled clinical trial conducted by the Malaria Vaccine and Drug Development Center (MVDC/CIV) in collaboration with ASOCLINIC IPS and the Pacific Health Institute (INSALPA) in Quibdó, Chocó, Colombia. A total of 72 healthy adults aged 18-50 years from malaria-endemic areas will participate.

Participants will be randomly assigned in a 2:1 ratio to receive either the PvCS/Montanide ISA-51 vaccine or a placebo. The study product will be administered by intramuscular injection at months 0, 2, and 4. After each vaccination, participants will be monitored for side effects and provide blood samples to measure immune responses, including antibody levels and T-cell activity.

Approximately one month after the third vaccination, participants will undergo a controlled human malaria infection (CHMI), during which they will be exposed to P. vivax through the bite of infected mosquitoes under strict medical supervision. Following exposure, participants will be monitored daily using blood tests to detect malaria at the earliest stage.

If malaria parasites are detected-or if 21 days pass without infection-participants will receive prompt, effective antimalarial treatment based on Colombian national guidelines. All participants will continue to be followed for up to 12 months after the challenge to ensure safety and assess long-term outcomes.

Primary goals of the study include:

Determining whether the PvCS/Montanide ISA-51 vaccine prevents P. vivax infection after CHMI.

Measuring the time between exposure and first detection of parasites (pre-patent period).

Evaluating the safety and tolerability of the vaccine.

Secondary goals include:

Measuring immune responses generated by the vaccine. Exploring relationships between immune responses and protection from infection. The total duration of the study is expected to be approximately 30 months, including recruitment, immunizations, challenge procedures, and follow-up. Results will help determine whether this vaccine can safely protect adults against P. vivax malaria and guide planning for future larger-scale vaccine trials in endemic populations.

DETAILED DESCRIPTION:
This Phase IIa/b randomized, double-blind, placebo-controlled clinical trial is designed to evaluate the protective efficacy, safety, and immunogenicity of the PvCS/Montanide ISA-51 vaccine when followed by a controlled human malaria infection (CHMI) with Plasmodium vivax. The investigational product consists of synthetic peptides representing the central repeat and flanking regions of the P. vivax circumsporozoite (CS) protein formulated with the Montanide ISA-51 adjuvant. This vaccine formulation was selected based on earlier phase studies demonstrating acceptable safety and immune reactivity in adults.

The study will enroll 72 healthy adults aged 18-50 years residing in a malaria-endemic region of Chocó, Colombia. Participants will be randomized in a 2:1 ratio to receive either the PvCS/Montanide ISA-51 vaccine or placebo. Vaccinations will be administered intramuscularly at months 0, 2, and 4. Safety assessments will include clinical evaluations, laboratory monitoring, and systematic documentation of all adverse events throughout the vaccination and follow-up periods.

Immunogenicity will be characterized using standardized assays to quantify antibody responses (ELISA and indirect immunofluorescence) and cellular responses (ELISpot), including measurements of IFN-γ-secreting T cells. Samples will be collected at predefined time points to evaluate the magnitude, kinetics, and durability of immune responses.

Approximately one month after the third vaccination, participants will undergo CHMI via exposure to Anopheles albimanus mosquitoes infected with P. vivax sporozoites. The challenge will be conducted in a controlled setting with continuous clinical oversight. After CHMI, participants will undergo daily parasitological monitoring by thick smear, supplemented by PCR assays, until the detection of parasitemia or for up to 21 days post-challenge.

Participants who develop parasitemia will receive immediate antimalarial treatment according to national guidelines. Extended follow-up will include evaluations of treatment response, late-onset adverse events, and persistence of vaccine-induced immune responses for up to 12 months after CHMI.

The primary objectives are to determine whether vaccination with PvCS/Montanide ISA-51 reduces the risk of developing P. vivax parasitemia after CHMI and whether it prolongs the pre-patent period compared with placebo. Safety outcomes include the frequency and severity of local, systemic, and laboratory adverse events. Secondary objectives include detailed characterization of humoral and cellular responses and exploratory analyses assessing associations between immunogenicity and protection.

The study is expected to last approximately 30 months, including recruitment, immunization, challenge procedures, and follow-up. Results will provide critical data to guide future development of P. vivax CS-based vaccines and inform decisions regarding advancement to larger efficacy trials in endemic settings.

.

ELIGIBILITY:
Inclusion Criteria Age 18-50 years, male or female. Healthy adults, as determined by medical history, physical examination, and screening laboratory tests.

Able and willing to provide written informed consent prior to any study procedure.

Available for the full duration of the study, including follow-up through 12 months post-challenge.

Group-specific criteria:

Malaria-naïve cohort: No prior malaria infection or residence in malaria-endemic areas; negative malaria serology at screening.

Semi-immune cohort: Residence ≥ 5 years in a P. vivax-endemic area and documented or self-reported prior malaria exposure.

Screening negative for HIV, hepatitis B surface antigen (HBsAg), and hepatitis C virus antibodies.

For women of childbearing potential:

Negative pregnancy test at screening and prior to each vaccination and/or CHMI. Commitment to use effective contraception (hormonal, IUD, barrier methods, or abstinence) from screening through the end of follow-up.

Willingness to comply with all study procedures, including repeated blood sampling, controlled human malaria infection (CHMI), and inpatient or outpatient monitoring as required.

Exclusion Criteria Previous participation in any malaria vaccine clinical trial or any controlled human malaria infection (CHMI) study.

History of severe allergic reactions, including anaphylaxis, to vaccines or vaccine components such as Montanide ISA-51 VG, adjuvants, or synthetic peptides.

Clinically significant acute or chronic medical conditions that may increase risk or interfere with study participation, including but not limited to:

Cardiovascular disease Hepatic or renal impairment Neurological or psychiatric disorders Autoimmune diseases Hematologic abnormalities Immunodeficiency or immunosuppressive conditions Use of immunosuppressive therapies, systemic corticosteroids, antimalarial medications, or other agents that may interfere with vaccine immune responses within 30 days prior to enrollment.

Receipt of immunoglobulins or blood products within 3 months prior to screening.

Pregnancy or breastfeeding at screening or planned pregnancy during the study period.

Participation in another clinical trial of an investigational product or device within 30 days prior to enrollment or planned participation during the study.

Any clinically significant abnormality on screening laboratories, ECG, or physical examination that, in the investigator's judgment, could:

Pose a safety risk, Confound study results, or Impair adherence to study procedures. Any condition or circumstance that, in the investigator's opinion, could compromise volunteer safety or the integrity of the trial.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2026-01-19 (Estimated); Primary Completion 2027-07-12 (Estimated); Study Completion 2028-06-12 (Estimated)

PRIMARY OUTCOMES:
Protective Efficacy Against P. vivax Infection After Controlled Human Malaria Infection (CHMI) | Day 7 to Day 28 post-challenge.
  Definition: Proportion of volunteers who develop P.vivax parasitemia following exposure to 2-4 infected Anopheles albimanus mosquitoes. Parasitemia will be assessed daily by thick blood smear (GG). PCR will be performed as a confirmatory assay but will not to be used for clinical decision-making. Unit of Measure: Number and percentage of infected participants.

SECONDARY OUTCOMES:
Incidence of Local Adverse Events at the Injection and Mosquito Bite Site Within 7 Days Post-Challenge | Within 7 days post-challenge
  Number of participants experiencing local adverse events (AEs), including pain, erythema, or swelling, at injection or mosquito bite sites following the challenge, assessed and graded according to FDA Toxicity Grading Scale criteria.
  Unit: Number of participants with local AEs.
Incidence of Systemic Adverse Events Within 7 Days After Completion of Antimalarial Treatment | Within 7 days post-challenge
  Number of participants experiencing local adverse events, including pain, erythema, or swelling, at injection or mosquito bite sites following the challenge, assessed and graded according to FDA Toxicity Grading Scale criteria.
  Unit: Number of participants with SAEs
Incidence of Serious Adverse Events From First Vaccination Through 12 Months Post-Challenge | From first vaccination through 12 months post-challenge
  Number of participants experiencing serious adverse events (SAEs), as defined by International Council for Harmonisations Good Clinical Practice (ICH-GCP) guidelines, from the first vaccination through 12 months after challenge.
  Unit: Number of participants with SAEs.
Incidence of Laboratory Abnormalities in Hematology and Clinical Chemistry From Baseline to Day 60 Post-Challenge | From baseline to Day 60 post-challenge
  Number of participants with abnormal hematology or clinical chemistry results, including liver and kidney function tests, graded according to FDA Toxicity Grading Scale criteria, from baseline through Day 60 post-challenge.
  Unit: Number of participants with abnormal laboratory results.
Incidence of Coagulation and Urinalysis Abnormalities From Baseline to Day 60 Post-Challenge | From baseline to Day 60 post-challenge
  Number of participants with abnormal coagulation parameters or urinalysis results, graded according to FDA Toxicity Grading Scale criteria, from baseline through Day 60 post-challenge.
  Unit: Number of participants

OTHER OUTCOMES:
Anti-Plasmodium vivax Circumsporozoite Protein IgG Antibody Titers Measured by ELISA | Day 0, Months 1, 2, 3, 6, 7, 8.
  Quantification of IgG antibody titers against N-terminal, repeat (R), and C-terminal regions of the Plasmodium vivax circumsporozoite protein (PvCSP) measured using enzyme-linked immunosorbent assay (ELISA).
  Unit: Antibody titer
Anti-sporozoite IgG Antibody Titers Measured by Indirect Fluorescent Antibody test (IFAT) | Day 0, Months 1, 2, 3, 6, 7, 8.
  Quantification of IgG antibody titers against Plasmodium vivax sporozoites measured using the indirect fluorescent antibody test (IFAT).
  Unit: Reciprocal Antibody titer, measured as the highest dilution showing fluorescence.
Interferon-Gamma-Producing T-cell Responses Measured by ELISpot Assay | Day 0, Month 3, Month 6.
  Quantification of interferon-gamma (IFN-γ)-producing T-cell responses measured by ELISpot assay following stimulation with Plasmodium vivax circumsporozoite protein peptides.
  Unit: Spot-forming cells per number of peripheral blood mononuclear cells (PBMCs)Measured as spot-forming cell (SFCs) per 10^6PBMCs.
Time to First Microscopically Detected Parasitemia After Controlled Human Malaria Infection | Days 7 to 28 post-challenge.
  Number of days from controlled human malaria infection (CHMI) to the first detection of parasitemia by positive thick blood smear.
  Unit: Days
Parasitemia Density at First Positive Thick Blood Smear After Controlled Human Malaria Infection | Days 7-28 post-challenge.
  Density of parasitemia expressed as the number of parasites per microliter of blood measured at the time of the first positive thick blood smear following controlled human malaria infection.
  Unit: Parasites/µL
Incidence of Malaria-Related Signs and Symptoms From Day 0 to Day 28 Post-Challenge | Days 0 to Day 28 post-challenge.
  Number of participants experiencing malaria-related clinical signs and symptoms during the post-challenge follow-up period.
  Unit: Number of participants
Severity of Malaria-Related Signs and Symptoms Graded by FDA Toxicity Criteria From Day 0 to Day 28 Post-Challenge | Day 0 to Day 28 post-challenge
  Maximum severity grade of malaria-related clinical signs and symptoms per participant, assessed and graded according to FDA Toxicity Grading Scale criteria.
  Unit: Toxicity grade

CONTACTS AND LOCATIONS:
Overall Officials: Myriam Arevalo, PhD, Study Director — Malaria Vaccine and Drug Development Center (MVDC)
Locations (1):
- Malaria Vaccine and Drug Development Center (MVDC), Cali, Valle del Cauca Department, Colombia

IPD SHARING:
Plan to Share IPD: Yes
Access to the data will be provided upon reasonable request to the corresponding investigator. Requests must include a research proposal and will be reviewed for scientific merit and ethical compliance. Data will be shared in a de-identified format.
Supporting Information: Study Protocol, SAP
Time Frame: De-identified individual participant data and supporting documentation will be available after publication of the primary results of the study. Data may be requested for a period of up to five years following publication.
Access Criteria: Access to de-identified individual participant data will be granted upon reasonable request to the corresponding investigator. Requests must include a research proposal and will be evaluated for scientific validity, ethical compliance, and consistency with participant consent. Approved users will receive access to de-identified data only, with no direct identifiers.
URL: https://caucaseco.org/

DOCUMENTS (4):
  • Study Protocol (2025-08-07): https://cdn.clinicaltrials.gov/large-docs/01/NCT07373301/Prot_000.pdf
  • Informed Consent Form: Informed consent HIV (2025-08-07): https://cdn.clinicaltrials.gov/large-docs/01/NCT07373301/ICF_001.pdf
  • Informed Consent Form: Informed Consent Secondary Use Samples (2025-08-07): https://cdn.clinicaltrials.gov/large-docs/01/NCT07373301/ICF_002.pdf
  • Informed Consent Form: Informed consent Immunization (2025-08-07): https://cdn.clinicaltrials.gov/large-docs/01/NCT07373301/ICF_003.pdf